CLINICAL TRIAL: NCT01159041
Title: Evaluation of Family Focused Treatment for Childhood Depression
Brief Title: Systems of Support Study for Childhood Depression
Acronym: SOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: University of California, Los Angeles (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Martha C. Tompson, Associate Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01MH082861 (NIH); R01MH082856-01A2 (NIH); R01MH082861-01A2 (NIH)
Record Dates: First submitted 2010-07-07; First posted 2010-07-09 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Depression
Keywords: Depression, children, adolescent, family
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family Focused Treatment (FFT) (Experimental): 15 session family-based treatment emphasizing improving relationship skills to combat depression symptoms and support recovery.
  Interventions: Behavioral: Family Focused Treatment (FFT)
- Individual Treatment (IP) (Active Comparator): 15 session individually-based treatment to assist children in understanding the causes of their symptoms.
  Interventions: Behavioral: Individual Treatment (IP)

INTERVENTIONS:
Behavioral: Family Focused Treatment (FFT) — FFT is designed to specifically address the developmental needs of school-aged children and their parents through an emphasis on fostering positive and supportive parent-child interactions that scaffold the development of a positive self, to help parents provide the child additional positive feedback on his/her developmentally appropriate achievements, and to enhance family and child coping. This treatment is conducted with the child and his/her parent(s) and includes education about depression, communication training, relationship enhancement, and problem-solving.
  Arms: Family Focused Treatment (FFT)
Behavioral: Individual Treatment (IP) — The goals of the treatment are to foster the therapeutic relationship, to provide a supportive and empathic setting where the child can come to better understand his/her emotions/feelings and address issues underlying current symptoms. Therapeutic goals will be addressed through reflection and clarification of feelings/emotions and understanding the child's perception of the context of depressed feelings.
  Arms: Individual Treatment (IP)

SUMMARY:
This study is designed to compare two treatments for depression in pre-adolescent (7-13 year old) children. A family-focused treatment will be compared to an individual child-focused treatment in this 14-week intervention.

DETAILED DESCRIPTION:
Childhood-onset depression is an impairing and often recurrent and persistent disorder that impacts current and later development resulting in high personal, social, and economic costs. Despite the costs of early-onset depression, the emphasis in current practice parameters on an initial course of psychosocial treatment, and extensive research on adolescent depression, we currently lack randomized controlled trials evaluating psychosocial treatments for children with depressive disorders.

The present proposal aims to address this gap in knowledge regarding optimal psychosocial treatment strategies for children suffering from depressive disorders. We propose a 2-site randomized controlled trial to evaluate the efficacy of Family Focused Treatment (FFT), as compared to an individual client-centered psychotherapy (IP) modeled after "usual" community care. FFT adopts an interpersonal model for understanding how depressive symptoms are maintained, emphasizes developing family skills/strategies for altering interpersonal processes, and works on building a family environment that supports recovery and enhances stress resistance and resilience. This approach may be particularly appropriate to the developmental needs of depressed children, given their dependence on parents, the potential of FFT to address the needs of multiple family members, and our data supporting benefits on depression, functioning, and other co-occurring symptoms.

The proposed project will enroll 140 children (ages 8-12) with depressive disorders. Children will be randomly assigned to receive a 14-week trial of either FFT or IP. At study entry, immediately post-treatment, and at a 9-month post-treatment follow-up all participants will undergo intensive evaluation of clinical state and psychosocial and family functioning.

ELIGIBILITY:
Inclusion Criteria:

* current Depressive Disorder
* ages 7-13 years
* living with at least one biological parent willing to participate

Exclusion Criteria:

* thought disturbance
* severe conduct disorders
* unstable on antidepressant medications
* continuation in current non-study treatment
* non-English speaking

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 134 (Actual)
Dates: Start 2010-01; Primary Completion 2015-05 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Adequate Depression Treatment Response | 3 months
  50% improvement on Children's Depression Rating Scale-Revised

SECONDARY OUTCOMES:
Interviewer-rated Depression Severity | 3 Months
  Children's Depression Rating Scale-Revised (CDRS-R) measures depression severity over the past two weeks. The 17-item CDRS-R has total scores ranging from 17 to 113 with scores of 40 or greater considered indicative of a depression diagnosis. Used in pharmacological and psychosocial treatment studies, it provides comparability across studies.
Children's Self-Report of Depression Symptoms | 3 Months
  Child Depression Inventory (CDI) is a 27-item self-report measure. Scores range from 0 to 54 with higher scores reflecting higher levels of symptoms.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UCLA Semel Institute for Neuroscience and Human Behavior, Los Angeles, California
  - Boston University, Boston, Massachusetts

REFERENCES:
- [Background] Tompson MC, Pierre CB, Haber FM, Fogler JM, Groff AR, Asarnow JR. Family-focused treatment for childhood-onset depressive disorders: results of an open trial. Clin Child Psychol Psychiatry. 2007 Jul;12(3):403-20. doi: 10.1177/1359104507078474. PMID 17953128
- [Result] Tompson MC, Boger KD, Asarnow JR. Enhancing the developmental appropriateness of treatment for depression in youth: integrating the family in treatment. Child Adolesc Psychiatr Clin N Am. 2012 Apr;21(2):345-84. doi: 10.1016/j.chc.2012.01.003. Epub 2012 Mar 17. PMID 22537731
- [Result] Tompson MC, Sugar CA, Langer DA, Asarnow JR. A Randomized Clinical Trial Comparing Family-Focused Treatment and Individual Supportive Therapy for Depression in Childhood and Early Adolescence. J Am Acad Child Adolesc Psychiatry. 2017 Jun;56(6):515-523. doi: 10.1016/j.jaac.2017.03.018. Epub 2017 Apr 7. PMID 28545757
- [Result] Tompson MC, Langer DA, Hughes JL, Asarnow JR. Family-Focused Treatment for Childhood Depression: Model and Case Illustrations. Cogn Behav Pract. 2017 Aug;24(3):269-287. doi: 10.1016/j.cbpra.2016.06.003. PMID 28966545
- [Derived] Asarnow JR, Tompson MC, Klomhaus AM, Babeva K, Langer DA, Sugar CA. Randomized controlled trial of family-focused treatment for child depression compared to individual psychotherapy: one-year outcomes. J Child Psychol Psychiatry. 2020 Jun;61(6):662-671. doi: 10.1111/jcpp.13162. Epub 2019 Dec 15. PMID 31840263